CLINICAL TRIAL: NCT03953950
Title: Effect of Add-on Spironolactone to Losartan Versus Losartan Alone on Peritoneal Membrane Among Continuous Ambulatory Peritoneal Dialysis Patients: An Open-Label Randomized-Controlled Trial
Brief Title: Effect of Add-on Spironolactone to Losartan Versus Losartan Alone on Peritoneal Membrane Among Peritoneal Dialysis Patients
Acronym: ESCAPE-PD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Chidchanok Ruengorn, Principal Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THOR Study Group
Record Dates: First submitted 2019-04-20; First posted 2019-05-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis
Keywords: Peritoneal Dialysis; Peritoneal Membrane; Spironolactone; Losartan; Renin-Angiotensin-Aldosterone System
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Spironolactone; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination of spironolactone and losartan (Experimental)
  Interventions: Drug: Spironolactone; Drug: Losartan
- Losartan Alone (Active Comparator)
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Spironolactone — Spironolactone Starting dose: 25 mg/day Target dose: 100 mg/day Titration: every 1-2 weeks, based on BP (keep< 140/90 mmHg, but avoid hypotension <90/60 mmHg), and serum potassium level (<5.5 milliequivalent /liter)
  Arms: Combination of spironolactone and losartan
Drug: Losartan — Losartan Starting dose: 50 mg/day Target dose: 100 mg/day Titration: every 1-2 weeks, based on BP (keep< 140/90 mmHg, but avoid hypotension <90/60 mmHg), and serum potassium level (<5.5 milliequivalent /liter)

SUMMARY:
The ESCAPE-PD (Effects of add-on SpironolaCtone to losartan versus Alone on Peritoneal mEmbrane among continuous ambulatory Peritoneal Dialysis patients) study is a randomized, open-label, single center, active-controlled clinical trial. Adults end-stage kidney disease patients 18 years or older undergoing continuous ambulatory peritoneal dialysis (CAPD) will be enrolled. A total 84 CAPD will be randomly assigned to either the combination of spironolactone and losartan (experimental arm) or losartan alone (control arm). The primary outcomes are the difference in peritoneal dialysate effluent cancer antigen-125 (CA-125) and peritoneal equilibration test (PET) indices (dialysate-to-plasma creatinine ratio, 4-hour ultrafiltration volume, and the concentration of glucose present in the solution at the start of the test). Secondary outcome measures include laboratory and mechanistic outcome measures, nutrition outcomes, health-related quality of life, physical function, clinical events, and safety profiles. Results will be disseminated to suggest a strategy to prevent the peritoneal membrane function among CAPD patients through peer-reviewed publications along with scientific meetings.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is one of the methods of renal replacement therapy (RRT) that can easily perform at home. The declared "PD first" policy from the National Health Security Office causes rapidly expansion of this group of patients. In the year 2013, the current study in Thailand showed that the patients enrolled for peritoneal dialysis accumulated for more than 15,000 people. It works continuously similar to the actual function of the kidneys in normal people. In addition, PD also helps to slow the decline of remaining kidney function (residual renal function), which is very important and affect in decreasing mortality rate in this group of patients. However, PD has several limitations such as complications from the infection and high failure rate associated with a dysfunction of the peritoneal membrane during long-term treatment. Approximately 4-12 percent of patients will have ultrafiltration failure and volume overload in the first couple of years of treatment and soar to 30-50 percent in patients treated for more than six years.

The causes of peritoneal membrane deterioration are exposure to incompatible dialysis solution with hyperosmolar glucose content, acidic pH, reactions to PD catheter material, uremia and peritonitis. The alterations of structural and functional of the peritoneal membrane after exposed to these several insults are epithelial-to-mesenchymal transition (EMT), and increase in peritoneal solute transport, which consequently leading to peritoneal dialysis failure. It has been already demonstrated that the local renin-angiotensin-aldosterone system (RAAS) plays a key role in this regulation by promoting the activation of neoangiogenesis and fibrotic pathways.

According to the pathophysiologic changes of the peritoneal membrane, Angiotensin Converting Enzyme Inhibitors (ACEIs) and Angiotensin Receptor Blockers (ARBs) are adapted to be use in respect of membrane preserving agents. Many studies, both in human and animal models, demonstrate the protective effect against peritoneal membrane deterioration by inhibiting the formation of transforming growth factor beta1 (TGF-β1), vascular endothelial growth factor (VEGF), and decreasing progression rate of small to high transport membrane type. In fact, mineralocorticoid receptor antagonists (MRAs) seem to have higher efficacy than ACEIs/ARBs in some experimental models. The possible mechanism is the effects of mineralocorticoid receptor antagonists that not only inhibit the formation of TGF- β1 and VEGF, but also suppress intracellular Reactive Oxygen Species (ROS) generation, activation of extracellular signal-regulated kinase (ERK) 1/2, and p38 mitogen-activated protein kinase (MAPK), the substrates responsible for aldosterone induces alterations in cell phenotype. A prospective cohort study of 23 CAPD patients was conducted and evaluated the effect of spironolactone on peritoneal membrane. The result showed the possible benefit of spironolactone in slowing the decline of peritoneal function, suppressing the elevation of profibrotic markers, and increasing mesothelial cell mass.

As a result of the clinical practice, most of CAPD patients tend to receive ACEIs/ARBs as prescribe by the clinicians, in order to control blood pressure, raise serum potassium level, and others compelling indications. Thus, the concept of add-on MRAs to ACEIs/ARBs, desiring the synergistic effects of these 2 drugs group, for membrane preservation is challenge. Notwithstanding the fact that current evidence about the combination effects of ACEIs/ARBs with MRAs is limited in term of quality of the study, sample size, inadequate follow-up period, and poor sensitive parameter in assessing the structural and functional changes of the peritoneal membrane. Thereby, this study aims to evaluate the effect of add-on spironolactone to losartan versus losartan alone on membrane preservation in continuous ambulatory peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older (both male and female patients)
* Incidence or prevalent end-stage kidney disease patients undergoing CAPD
* Had standard dialysis prescription for at least 30 days before screening
* History of hypertension
* Stable clinical condition without any inflammation at least 4 weeks prior to enrolment
* Had an ability to understand and willingness to sign an informed consent statement

Exclusion Criteria:

* Serum potassium concentration of ≥ 5.5 milliequivalent /liter
* History of severe or active cardiovascular and/or cerebrovascular disease
* History of renal artery stenosis
* Uncontrolled hypertension
* Contraindication to angiotensin-converting enzyme inhibitors/angiotensin II receptor blockers or mineralocorticoid receptor antagonists
* Pregnancy
* Recent PD-related peritonitis or exit-site and tunnel infection (within 2 months of screening)
* Had planned to have kidney transplantation or transfer to other PD centers with 6 months
* Prognosis for survival less than 12 months
* Any conditions (both mental or physical) that would interfere with the participant's ability to comply with the study protocol
* Any disease of the abdominal wall, such as injury or surgery, burns, hernia, dermatitis, inflammatory bowel diseases (Crohn's disease, ulcerative colitis or diverticulitis) that in the opinion of the Investigator would preclude the patient from being able to have PD
* Any intra-abdominal tumors or intestinal obstruction
* Current or recent (within 30 days) exposure to others investigational medicinal products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Peritoneal dialysate effluent CA-125 | 6 months
  Using a commercial microparticle enzyme-linked immunosorbent assay
PET indices | 6 months
  PET indices including dialysate-to-plasma creatinine ratio [D/P Cr], 4-hour ultrafiltration (UF) volume, and the concentration of glucose present in the solution at the start of the test [D/D0]) measured using a modified PET method (performed using 2,000 mL of 2.5% glucose solution).

SECONDARY OUTCOMES:
Changes in dialysate adequacy by Weekly kt/V | 6 months
Changes in dialysate adequacy by weekly creatinine clearance | 6 months
Changes in serum albumin concentration | 6 months
Changes in serum potassium concentration | 6 months
Changes in waist circumference | 6 months
Changes in body mass index (BMI) | 6 months
  Weight and height will be combined to report BMI in kg/m^2
Changes in Nutritional status | 6 months
  Using Subjective Global Assessment (SGA)
Changes in Malnutrition-Inflammation Score (MIS) | 6 months
Changes in participant quality of life score | 6 months
  Using Kidney Disease Quality of Life-36 (KDQOL-36 Version 1.3)
Changes in health utility | 6 months
  Using EuroQOL-5 dimension 5-level (EQ-5D-5L)
Changes in disease-specific Thai quality of life score | 6 months
  Using the 9-Thai Health status AssessmentInstrument (9-THAI) questionnaire
Changes in participant well-being score | 6 months
  Using the World Health Organization-Five (WHO-5) well-being index
Number of participants with disability | 6 months
  Using the Barthel activities daily life index

OTHER OUTCOMES:
Changes in blood pressure | 6 months
Incidence of PD technique failure | 6 months
Incidence of PD-related infections | 6 months
  Peritonitis or exit-site and tunnel infection
Number of participants with investigational medicinal products-related adverse events as assessed by CTCAE v4.0 | 6 months
  Safety of investigational medicinal products related to potential harm (e.g. death, hospitalization, and emergency visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacoepidemiology and Statistics Research Center, Faculty of Pharmacy, Chiang Mai University, Chiang Mai, Thailand

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138